CLINICAL TRIAL: NCT04395716
Title: A Phase I Study of ResCure™ to Treat COVID-19 Infection
Brief Title: A Study of ResCure™ to Treat COVID-19 Infection
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Not ever started
Sponsor: ProgenaBiome (Other)
Collaborators: Rinati Skin, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRG-048
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: COVID; Covid-19; Corona Virus Infection; Sars-CoV2; Coronavirus-19; SARS Pneumonia; SARS-Associated Coronavirus as Cause of Disease Classified Elsewhere
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): This group will be treated with nebullized ResCure™ while hospitalized every 4 to 6 hours, depending on disease severity and ventilator status.
  Interventions: Biological: ResCure™

INTERVENTIONS:
Biological: ResCure™ — Patients will be treated with nebulized ResCure™

SUMMARY:
This is a Phase I open-label interventional study which will test the efficacy of ResCure™ in the treatment of patients with COVID-19 infection.

DETAILED DESCRIPTION:
In this Phase I open-label interventional study we will test the efficacy of ResCure™ in the treatment of patients with COVID-19 infection. Patients being treated will have severe respiratory symptoms that are at or near requiring the patient be placed on a ventilator.

ELIGIBILITY:
Inclusion Criteria:

1. Critically ill patients with SARS from COVID-19 infection on respirators OR
2. Patients with SARS from COVID-19 infection prior or after being placed on respirator
3. Male or female patients 18 years of age and older

Exclusion Criteria:

1. Patients less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
The rate of recovery of mild or moderate COVID-19 in patients using ResCure™ | 12 Weeks
  Number of days from COVID-19 diagnosis to recovery via RT-PCR
Reduction or progression of symptomatic days | 12 Weeks
  Reduction and/or progression of symptomatic days, reduction of symptom severity
Assess the safety of ResCure™ via pulse | 12 Weeks
  Pulse from baseline to 12 weeks
Assess the safety of ResCure™ via oxygen saturation | 12 Weeks
  Oxygen saturation from baseline to 12 weeks
Assess the safety of ResCure™ via EKG | 12 Weeks
  EKG from baseline to 12 weeks
Assess Tolerability of ResCure™ | 12 Weeks
  Assess Adverse Events and Serious Adverse Events due to ResCure™

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Principal Investigator — ProgenaBiome
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No